CLINICAL TRIAL: NCT01014390
Title: A Multi-Center, Prospective Study of the WallFlex Biliary RX Fully Covered Stent for the Treatment of Benign Biliary Strictures
Brief Title: WallFlex Biliary Fully Covered (FC) Benign Stricture Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDM 00027550
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Biliary Stricture
Keywords: benign biliary strictures secondary to chronic pancreatitis/post abdominal surgery/post liver transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WallFlex Biliary RX FC Stent System (Experimental): The WallFlex Biliary RX Fully Covered Stent System is being evaluated for treatment of benign biliary strictures.
  Interventions: Device: WallFlex Biliary RX Fully Covered Stent System

INTERVENTIONS:
Device: WallFlex Biliary RX Fully Covered Stent System — Temporary placement of a biliary stent as a treatment of biliary obstruction resulting from benign bile duct strictures. The stent is fully covered with a silicone polymer to reduce the potential of tissue ingrowth into the stent. The stent is removed after 5 months (±1 month) after stent placement in Post-Liver Transplant patients and after 11 months (±1 month) in Chronic Pancreatitis and Post-Abdominal Surgery patients.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the WallFlex® Biliary RX Fully Covered Stent as a treatment of biliary obstruction resulting from benign bile duct strictures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study
* Chronic pancreatitis or prior liver transplantation or prior other abdominal surgery (to include cholecystectomy)
* Indicated for ERCP procedure with stent placement for: Symptomatic bile duct stricture (i.e. obstructive jaundice, persistent cholestasis, acute cholangitis) confirmed by cholangiogram and/or Bile duct stricture confirmed by cholangiogram and/or Exchange of prior plastic stent(s) for management of benign stricture

Exclusion Criteria:

General:

* Placement of the stent in strictures that cannot be dilated enough to pass the delivery system
* Placement of the stent in a perforated duct
* Placement of the stent in very small intrahepatic ducts
* Patients for whom endoscopic techniques are contraindicated
* Biliary stricture of malignant etiology
* Biliary stricture of benign etiology other than chronic pancreatitis or liver transplant anastomosis or other abdominal surgery
* Stricture within 2 cm of duct bifurcation
* Symptomatic duodenal stenosis (with gastric stasis)
* Prior biliary self-expanding metal stent
* Suspected stricture ischemia based on imaging of hepatic artery occlusion or endoscopic evidence of biliary cast syndrome
* Known bile duct fistula
* Known sensitivity to any components of the stent or delivery system
* Participation in another investigational study within 90 days prior to consent or during the study

Additional Specific to Chronic Pancreatitis Patients:

* Developing obstructive biliary symptoms associated with an attack of acute pancreatitis

Additional Specific to Post-Abdominal Surgery Patients:

* History of hepatectomy
* History of liver transplant

Additional Specific to Liver Transplant Patients:

* Live donor transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Westmead Hospital, Westmead, New South Wales, Australia
- Medical University of Vienna, Vienna, Austria
- ULB Erasme Hospital, Brussels, Belgium
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal-Saint-Luc Hospital, Montreal, Quebec
  - MUHC - McGill University, Montreal, Quebec
- Clinica Alemana de Santiago, Santiago, Chile
- Hopital Edouard Herriot, Lyon, France
- Evangelischen Krankenhaus, Düsseldorf, Germany
- Asian Institute of Gastroenterology, Hyderabad, India
- Università Cattolica del Sacro Cuore Policlinico A. Gemelli, Rome, Italy
- Erasmus Medical Center, Rotterdam, Netherlands
- Hospital Universitari Doctor Josep Trueta, Girona, Catalonia, Spain

REFERENCES:
- [Result] Deviere J, Nageshwar Reddy D, Puspok A, Ponchon T, Bruno MJ, Bourke MJ, Neuhaus H, Roy A, Gonzalez-Huix Llado F, Barkun AN, Kortan PP, Navarrete C, Peetermans J, Blero D, Lakhtakia S, Dolak W, Lepilliez V, Poley JW, Tringali A, Costamagna G; Benign Biliary Stenoses Working Group. Successful management of benign biliary strictures with fully covered self-expanding metal stents. Gastroenterology. 2014 Aug;147(2):385-95; quiz e15. doi: 10.1053/j.gastro.2014.04.043. Epub 2014 May 4. PMID 24801350
- [Derived] Poley JW, Ponchon T, Puespoek A, Bruno M, Roy A, Peetermans J, Rousseau M, Lepilliez V, Dolak W, Tringali A, Blero D, Carr-Locke D, Costamagna G, Deviere J; Benign Biliary Stenoses Working Group. Fully covered self-expanding metal stents for benign biliary stricture after orthotopic liver transplant: 5-year outcomes. Gastrointest Endosc. 2020 Dec;92(6):1216-1224. doi: 10.1016/j.gie.2020.04.078. Epub 2020 May 15. PMID 32417298
- [Derived] Tringali A, Reddy DN, Ponchon T, Neuhaus H, Llado FG, Navarrete C, Bruno MJ, Kortan PP, Lakhtakia S, Peetermans J, Rousseau M, Carr-Locke D, Deviere J, Costamagna G; Benign Biliary Stenoses Working Group. Treatment of post-cholecystectomy biliary strictures with fully-covered self-expanding metal stents - results after 5 years of follow-up. BMC Gastroenterol. 2019 Dec 12;19(1):214. doi: 10.1186/s12876-019-1129-3. PMID 31830897
- [Derived] Lakhtakia S, Reddy N, Dolak W, Ponchon T, Bruno MJ, Bourke MJ, Neuhaus H, Roy A, Gonzalez-Huix Llado F, Kortan PP, Peetermans J, Rousseau M, Costamagna G, Deviere J; Benign Biliary Stenoses Working Group. Long-term outcomes after temporary placement of a self-expanding fully covered metal stent for benign biliary strictures secondary to chronic pancreatitis. Gastrointest Endosc. 2020 Feb;91(2):361-369.e3. doi: 10.1016/j.gie.2019.08.037. Epub 2019 Sep 5. PMID 31494135
- See also: Successful management of benign biliary strictures with fully covered self-expanding metal stents. — http://www.ncbi.nlm.nih.gov/pubmed/?term=24801350

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WallFlex Biliary RX FC Stent System
Started | 187
Completed | 177
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | WallFlex Biliary RX FC Stent System
Number analyzed (Participants) | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 168
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 145
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 18
  Netherlands | 17
  Austria | 24
  Belgium | 27
  Italy | 15
  France | 22
  Australia | 10
  Chile | 3
  Germany | 10
  India | 34
  Spain | 7

OUTCOME MEASURES:

1. Primary Outcome: Stent Removability
Description: Defined as ability to remove the stent endoscopically without serious stent removal related adverse events as assessed from the time of stent removal to 1month post-stent removal.
Time Frame: At stent removal
Population: 10 Patients were excluded because of death (from unrelated cause), withdrawal of consent, or switch to palliative treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Biliary RX FC Stent System
Number analyzed (Participants) | 177
Participants | 132

ADVERSE EVENTS:
Groups:
- WallFlex Biliary RX FC Stent System: evaluated for treatment of benign biliary strictures.
Arm/Group | WallFlex Biliary RX FC Stent System
Serious Adverse Events (participants affected / at risk) | 51/187
Other Adverse Events (participants affected / at risk) | 0/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WallFlex Biliary RX FC Stent System (N=187)
Cholangitis/fever (Gastrointestinal disorders) | 26
Abdominal pain (Gastrointestinal disorders) | 10
Pancreatitis (Gastrointestinal disorders) | 5
Cholecystitis (Gastrointestinal disorders) | 3
Cholestasis (Gastrointestinal disorders) | 3
Other (Gastrointestinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No